CLINICAL TRIAL: NCT03776643
Title: Safety and Efficacy of Low-dose IL-2 in Birch Pollen Allergy
Acronym: Rhinil-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160936J
Record Dates: First submitted 2018-11-20; First posted 2018-12-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-12

CONDITIONS: Allergic Rhinoconjunctivitis to Birch Pollen; With a Positive Skin Prick Test to Birch Pollen

STUDY DESIGN:
Intervention Model Description: Safety/Efficacy
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILT-101 (ld-IL2) (Experimental): Subcutaneous injections of ILT-101
  Interventions: Drug: ILT-101 ld-(IL2)
- placebo (Placebo Comparator): Subcutaneous injections of placebo
  Interventions: Drug: ILT-101 ld-(IL2)

INTERVENTIONS:
Drug: ILT-101 ld-(IL2) — Subcutaneous injections of ILT-101 or Placebo starting with once-daily administration for 5 consecutive days followed by once every two weeks administration during five months
  Other Names: Placebo

SUMMARY:
Several studies have reported a deficit and/or a defect in regulatory T cells in allergic subjects, which can be correlated with the allergic responses, especially for respiratory allergies. Low-dose IL-2 (ld-IL2) specifically targets and activates regulatory T cells (Tregs), which are cells that regulate immune responses. Thus by stimulating Tregs, ld-IL2 would control allergic responses.

This study is designed to evaluate the efficacy of ILT-101 (ld-IL-2), compared to placebo, on the nasal response assessed by Total Nasal Symptom Score (TNSS) during a controlled birch allergen exposure.

DETAILED DESCRIPTION:
Primary objective To evaluate the efficacy of ILT-101 (ld-IL-2), compared to placebo, on nasal response on day 40

Secondary objectives To evaluate the efficacy of ILT-101 on rhino-conjunctivitis symptoms, on inflammatory mediators, allergic specific immune responses and safety.

Experimental design This is a monocentric, randomized, placebo controlled, double-blind trial in parallel-groups, evaluating a treatment by ILT-101/placebo, 1 MIU daily for 5 days and 1 MIU every week, until day 36.

Population involved Male or female, aged between 18 and 55 years, with allergic rhinitis to birch pollen.

Number of subjects: 24

Duration of patient participation: 3 months (treatment period: 36 days months, follow-up period: 34 days)

ELIGIBILITY:
Inclusion criteria

* male or female aged between18-55 years
* Positive clinical history of seasonal allergic rhinitis to birch pollen for at least 2 consecutive pollinic seasons before inclusion and requiring medication intake with or without GINA 1 associated asthma, with documentation of sensitivity within 12 months before enrollment by : *Positive skin prick test (SPT) and validated in vitro tests for specific Immunoglobulin E (IgE); *Positive Skin prick test (SPT): wheal for birch pollen ≥ 5 mm in diameter for histamine wheal ≥ 3 mm (positive control) and NaCl reaction < 2 mm (negative control) *Positive specific IgE to birch pollen >0.75 kUI/L;
* Negative beta-HcG pregnancy test at screening visit for women of childbearing age;
* Normal electrocardiogram without clinically significant abnormalities;
* Ability to stay in the EEC for up to 4 hours, without any conditions or factors which could make this not possible
* Positive nasal response (TNSS≥5) at baseline exposure
* Free, informed and written consent signed by the patient and the investigator, before any specific examination required by the study;
* Affiliation to a social security scheme (beneficiary or assignee)
* Negative SARS-CoV-2 test less than 72 hours prior to screening visit

Exclusion Criteria:

* Asthma: GINA 2 to 5
* Eosinophilia > 0.6x109/mL;
* Any history of anaphylactic reactions;
* Specific immunotherapy treatment at the moment, including Omalizumab;
* Specific immunotherapy for birch-pollens within 3 previous years;
* Use of systemic corticosteroid or others immunosuppressive treatment within previous 6 months;
* Moderate to severe allergic rhinoconjunctivitis with or without asthma due to grass pollen, if the study is performed during grass pollen season (according to ARIA)
* Significant rhinitis, or sinusitis, due to daily contact with other allergen causing symptoms that are expected to coincide with exposures, as assessed by the investigator
* Contraindications known to treatment with IL-2:

  * Hypersensitivity to the active substance or to any of the excipients;
  * Immunosuppressed patient;
  * Psychotropic, hepatotoxic, nephrotoxic, myelotoxic or cardiotoxic drugs;
  * Other chronic diseases not clinically controlled;
  * Signs of active infection requiring treatment;
  * Previous history of organ transplantation.
  * Heart failure (≥ grade II, class. NYHA), kidney failure (Cockroft <60 ml/min/1.73m2), liver failure (transaminase> 3N), pulmonary insufficiency (any grade);
* Leukocytes <3000 / mm3 lymphocytes <800 / mm3, platelets <80 000 / mm3, Hemoglobin < 10.0 g/dL or 6.2 mmol/L, red cell blood < 3.5 T/L;
* Positivity of at least one of the thyroid-specific antibodies (anti-TPO, anti-TG, or anti-TRAKS) associated with an abnormal thyroid workup (TSH, T3, or T4) at inclusion;
* Chronic uncontrolled arterial hypertension (Systolic BP > 140 mmHg and/or Diastolic BP > 90 mmHg);
* Poor venous capital will forbid blood samples;
* Vaccination with attenuated live vaccine in the month before the inclusion or planned during the study;
* Vaccination against COVID-19 during the study period or if the 2nd dose of vaccine is planned during the 15 days preceding Visit 3
* Surgery in the previous three months or anticipated under study;
* Participation in other interventional research with study drug in the previous month and during the study;
* Psychiatric illness or any other concomitant chronic illness or addiction that could interfere with the ability to meet the requirements of the protocol or provide informed consent;
* Presence or history of unhealed cancer for more than five years, presence or history of healed cancer for less than five years, except carcinoma in situ of the cervix or basal cell carcinoma;
* Pregnant or lactating women;
* Men and women of childbearing age without effective contraception during the treatment period;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Change in nasal congestion expressed as area under the curve (AUC), during birch allergen exposure in ALYATEC's Environmental Exposure Chamber (EEC) | on day 40
  Change in nasal congestion expressed as area under the curve (AUC), during birch allergen exposure in ALYATEC's Environmental Exposure Chamber (EEC)

SECONDARY OUTCOMES:
Change in nasal congestion expressed as area under the curve (AUC), assessed during 4 hours of exposure | at Day 8
  TNSS, expressed as area under the curve (AUC), assessed during 4 hours of exposure: TOTAL NASAL SYMPTOM SCORE Definition of response choices (drop down menu for each of the 4 questions below) 0 = None 1 = Mild (symptom clearly present but easily tolerated) 2 = Moderate (annoying but tolerable symptom) 3 = Severe (difficult to tolerate symptom, disrupts activities)
Change in nasal response intensity | at Day 8
  determined by Visual Analogue Scale (VAS) ranged from 0 to 10 cm where higher values correspond to more intense symptoms
Changes in Tregs expressed in percentag (%) | at day 8
  Changes in Tregs in percentag compared to baseline
Changes in Tregs expressed in percentag (%) | at day 40
  Changes in Tregs in percentag compared to baseline
Changes in Tregs expressed in percentag (%) | at day 70
  Changes in Tregs in percentag compared to baseline
Changes in absolute count in Tregs | at day 8
  Changes in absolute count in Tregs compared to baseline
Changes in absolute count in Tregs | at day 40
  Changes in absolute count in Tregs compared to baseline
Changes in absolute count in Tregs | at day 70
  Changes in absolute count in Tregs compared to baseline
Changes in eosinophils expressed in percentag (%) | at day 8
  Changes in eosinophils in percentag compared to baseline
Changes in eosinophils expressed in percentag (%) | at day 40
  Changes in eosinophils in percentag compared to baseline
Changes in eosinophils expressed in percentag (%) | at day 70
  Changes in eosinophils in percentag compared to baseline
Changes in absolute count in eosinophils | at day 8
  Changes in absolute count in eosinophils compared to baseline
Changes in absolute count in eosinophils | at day 40
  Changes in absolute count in eosinophils compared to baseline
Changes in absolute count in eosinophils | at day 70
  Changes in absolute count in eosinophils compared to baseline
Changes in Inate Lymphoid Cell type 2(ILC2) expressed in percentag (%) | at day 8
  Changes in Inate Lymphoid Cell type 2 in percentag compared to baseline
Changes in Inate Lymphoid Cell type 2(ILC2) expressed in percentag (%) | at day 40
  Changes in Inate Lymphoid Cell type 2 in percentag compared to baseline
Changes in Inate Lymphoid Cell type 2(ILC2) expressed in percentag (%) | at day 70
  Changes in Inate Lymphoid Cell type 2 in percentag compared to baseline
Changes in absolute count in Inate Lymphoid Cell type 2(ILC2) | at day 8
  Changes (in absolute count in Inate Lymphoid Cell type 2 compared to baseline
Changes in absolute count in Inate Lymphoid Cell type 2(ILC2) | at day 40
  Changes (in absolute count in Inate Lymphoid Cell type 2 compared to baseline
Changes in absolute count in Inate Lymphoid Cell type 2(ILC2) | at day 70
  Changes (in absolute count in Inate Lymphoid Cell type 2 compared to baseline
Changes of antigen-specific T-cell immune responses (cytokine IL-4 ) | at day 40
  cytokine IL-4 at day 40
Changes of antigen-specific T-cell immune responses (cytokine IL-4 ) | at day 70
  cytokine IL-4 at day 70
Changes of antigen-specific T-cell immune responses (cytokine IL-5) | at day 40
  cytokine IL-5 at day 40
Changes of antigen-specific T-cell immune responses (cytokine IL-5) | at day 70
  cytokine IL-5 at day 70
Changes of antigen-specific T-cell immune responses | at day 40
  IL-13 secretion after antigen restimulation at day 40
Changes of antigen-specific T-cell immune responses | at day 70
  IL-13 secretion after antigen restimulation at day 70
Changes in allergen-specific IgE dosages basophil activation test with pollen allergen | at day 40
  allergen-specific IgE dosages at day 40
Incidence of adverse events at day 8 | up to Day 8
  Adverse events throughout the study (according to NCI-CTC AE classification)
Incidence of adverse events at day 40 | up to Day 40
  Adverse events throughout the study (according to NCI-CTC AE classification)
Incidence of adverse events at 70 | up to Day 70
  Adverse events throughout the study (according to NCI-CTC AE classification)

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, Pr, Study Chair — APHP / CIC BTI / Hopital Pitie Salpétrière, Paris
Locations (2):
- France (2):
  - Centre d'essais cliniques, ALYATEC, Strasbourg, Environmental Exposure Chamber, Alyatec, 1 Place de L'hôpital
  - CIC Biothérapies - Service de Biothérapies, Paris, Groupe Hospitalier Pitié-Salpêtrière 47 -83 BD de L'hopital